CLINICAL TRIAL: NCT06897709
Title: "Stump-First" Approach in Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Orhan Üreyen, Asosc. prof, Izmir City Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10/05/2023, numbered 2023/61
Record Dates: First submitted 2025-02-05; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Acute Appendicitis; Acute Appendicitis with Appendix Abscess
Keywords: appendectomy; laparoscopic appendectomy; surgical tecnic
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: underwent laparoscopic appendectomy using the standard approach (Active Comparator): In Group 1, as part of the standard approach, the mesoappendix was initially ligated using LigaSure. After visualizing the base of the appendix, two hemoclips were applied on the stump side and one hemoclip on the appendix side. The tissue between was then divided with scissors, and the appendix was removed from the abdomen through the trocar in the umbilicus within an endobag.
  Interventions: Procedure: Classic Approach in Laparoscopic Appendectomy
- Group 2 underwent laparoscopic appendectomy using the Stump-First Approach (Active Comparator): Group 2, the cecal appendix was identified, and a window was created at the base of the appendix between the mesoappendix and the appendiceal wall. Two hemoclips were applied on the stump side, and one hemoclip on the appendix side. The tissue between was then divided with scissors. Finally, the mesoappendix was divided using LigaSure and the appendix was removed from the abdomen through the trocar in the umbilicus within an endobag
  Interventions: Procedure: Stump first Approach in Laparoscopic Appendectomy

INTERVENTIONS:
Procedure: Classic Approach in Laparoscopic Appendectomy — underwent laparoscopic appendectomy using the standard approach
  Arms: Group 1: underwent laparoscopic appendectomy using the standard approach
Procedure: Stump first Approach in Laparoscopic Appendectomy — Stump first Approach in Laparoscopic Appendectomy
  Arms: Group 2 underwent laparoscopic appendectomy using the Stump-First Approach

SUMMARY:
Objective: This study aims to compare the standard laparoscopic appendectomy with the "Stump-First Approach" technique in patients diagnosed with acute appendicitis in terms of intraoperative and postoperative complications that may occur (injury, intra-abdominal abscess, postoperative fever, and infection parameters).

DETAILED DESCRIPTION:
The patients were randomly assigned to two groups: Group 1 underwent laparoscopic appendectomy using the standard approach, and Group 2 underwent laparoscopic appendectomy using the Stump-First Approach. Randomization was performed using a specialized computer program. Pregnant women, individuals under 18 years of age, incidental appendectomies, patients with a history of plastron appendicitis, those with malignant pathology results, patients with additional pathologies aside from appendicitis, and those who underwent conventional appendectomy were excluded from the study. All operations were performed under general anesthesia. A single dose of cefazolin (2g, intravenous) was routinely administered as prophylactic antibiotic therapy during anesthesia induction. All surgeries were conducted under the supervision of a surgical specialist with at least five years of experience.

Surgical Technique: For both groups, access to the abdomen was achieved from below the umbilicus, through the use of a Veress needle for patients with no prior abdominal surgery, and through the Hasson technique for those with a history of abdominal surgery; establishing pneumoperitoneum, the abdomen was inserted with an initial 10 mm trocar. Under direct vision with a 30-degree optical aid, a 5 mm trocar was placed in the suprapubic region and a 10mm trocar in the left lower quadrant. The operating table was positioned at 15-20° Trendelenburg and 10-15° left lateral tilt.

In Group 1, as part of the standard approach, the mesoappendix was initially ligated using LigaSure. After visualizing the base of the appendix, two hemoclips were applied on the stump side and one hemoclip on the appendix side. The tissue between was then divided with scissors, and the appendix was removed from the abdomen through the trocar in the umbilicus within an endobag.

For Group 2, the cecal appendix was identified, and a window was created at the base of the appendix between the mesoappendix and the appendiceal wall. Two hemoclips were applied on the stump side, and one hemoclip on the appendix side. The tissue between was then divided with scissors. Finally, the mesoappendix was divided using LigaSure and the appendix was removed from the abdomen through the trocar in the umbilicus within an endobag. In both groups, the 10 mm trocar insertion site fascia was closed with 0 polyglactin and the skin with 3/0 polypropylene.

The groups were compared in infection status (white blood cell (WBC) count, C-reactive protein (CRP) levels, proportional changes in these parameters, additional antibiotic requirements). The sample size for the study was calculated using the G*Power 3.1 statistical power analysis program. Assuming α=0.05, power (1-β)=0.95, the case-intervention group allocation ratio 1:1, and a high effect size (Cohen's d=0.97) with a two-tailed analysis, the required sample size was determined to be 60 patients, with 30 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Acute appendicitis

Exclusion Criteria:

* exist of pregnancy, exist of cancer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The number of participants compared in infection status | 1 year
  The groups were compared in infection status (WBC, CRP, additional antibiotic requirements)

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No